CLINICAL TRIAL: NCT06277245
Title: A Phase 3 Randomized, Placebo-Controlled, Double-Blind Study to Evaluate LNK01001 in Adults Subjects With Moderate to Severe Atopic Dermatitis.
Brief Title: A Phase 3 Study of LNK01001 Capsule in Subjects With Moderate to Severe Atopic Dermatitis.
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Lynk Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LK001303
Record Dates: First submitted 2024-02-02; First posted 2024-02-26 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- LNK01001 12 mg (Experimental): o Period 1: Participants receive LNK01001 12 mg twice daily for 16 weeks. Period 2: Participants will continue on LNK01001 12 mg twice daily from Week 16 to Week 52.
  Interventions: Drug: LNK01001
- LNK01001 24 mg (Experimental): o Period 1: Participants receive LNK01001 24 mg twice daily for 16 weeks. Period 2: Participants will continue on LNK01001 24 mg twice daily from Week 16 to Week 52.
  Interventions: Drug: LNK01001
- Placebo / LNK01001 12 mg (Placebo Comparator): o Period 1: Participants receive a placebo twice daily for 16 weeks. Period 2: Participants will switch to receive LNK01001 12 mg twice daily from Week 16 to Week 52.
  Interventions: Drug: LNK01001; Drug: Placebo
- Placebo / LNK01001 24mg (Placebo Comparator): o Period 1: Participants receive a placebo twice daily for 16 weeks. Period 2: Participants will switch to receive LNK01001 24 mg twice daily from Week 16 to Week 52.
  Interventions: Drug: LNK01001; Drug: Placebo

INTERVENTIONS:
Drug: LNK01001 — Capsule; Oral
Drug: Placebo — Capsule; Oral
  Arms: Placebo / LNK01001 12 mg; Placebo / LNK01001 24mg

SUMMARY:
This is a randomized, double-blind study comparing LNK01001 to placebo in participants with moderately to severely atopic dermatitis who were candidates for systemic therapy (ie, patients with a history of inadequate response to topical treatments, those who were using a systemic treatment, or those for whom topical treatments are otherwise medically inadvisable).

The objective of this study is to evaluate the efficacy and safety of LNK01001 in adult patients with moderate to severe AD who are candidates for systemic therapy.

DETAILED DESCRIPTION:
This study includes a 35-day screening period; a 16-week randomized, placebo-controlled treatment period (Period 1); a 36-week long-term extension period (Period 2); and a 28 to 35-day follow-up period (FU).

Participants who meet eligibility criteria will be randomized in a 2:2:1:1 ratio to four treatment groups:

Group 1: LNK01001 12 mg BID (Day 1 to Week 16)， LNK01001 12 mg BID (Week 16 and thereafter) Group 2: LNK01001 24 mg BID (Day 1 to Week 16)， LNK01001 24 mg BID (Week 16 and thereafter) Group 3: Placebo (Day 1 to Week 16)， LNK01001 12 mg BID (Week 16 and thereafter) Group 4: Placebo (Day 1 to Week 16)， LNK01001 24 mg BID (Week 16 and thereafter)

Starting at Week 4, rescue therapy is allowed if medically necessary and the following parameters are met:

At Week 4 through Week 24: subjects with < 50% reduction in EASI response at any two consecutive scheduled visits, compared to the Baseline EASI score.

After Week 24: subjects with < 50% reduction in EASI at any scheduled or unscheduled visit, compared to the Baseline EASI score.

Starting at Week 16, the use of any concomitant topical medication for atopic dermatitis can be administered per the investigator's discretion and will no longer be considered as rescue therapy for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least ≥18 and ≤75 years of age.
* The subject has a diagnosis of atopic dermatitis for at least 1 year.
* Meets the following disease activity criteria: BSA ≥10% of AD involvement. EASI ≥16. IGA ≥3. WI-NRS ≥4.
* Documented history of inadequate response to topical corticosteroids (TCS) or topical calcineurin inhibitor (TCI) or documented systemic treatment for AD within 6 months before Baseline Visit.

Exclusion Criteria:

* Vaccinated or exposed to a live or attenuated vaccine within the 6 weeks prior to the first dose of investigational product unable or unwilling to discontinue current atopic dermatitis treatments before the study.
* Requirement of prohibited medications during the study.
* Other active skin diseases or skin infections requiring systemic treatment or would interfere with appropriate assessment of atopic dermatitis lesions.
* History of malignancy or current diagnosis of malignancy before screening visit.

In the opinion of the investigator or sponsor, any uncontrolled clinically significant laboratory abnormality that would affect the interpretation of study data or the subject's participation in the study uncontrolled diabetes, hypertension, kidney disease, liver disease, or severe heart disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Estimated)
Dates: Start 2024-02-06 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Eczema Area and Severity Index (EASI-75) at Week 16 | Baseline and Week 16
  EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness (erythema, inflammation), thickness (induration, papulation, swelling - acute eczema), scratching (excoriation), and lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease .
Investigator's Global Assessment (IGA) score of 0/1 at Week 16 | Baseline and Week 16
  Proportion of subjects achieving Investigator's Global Assessment (IGA) score of clear (0) or almost clear (1) and a reduction from baseline of ≥2 points at Week 16.

SECONDARY OUTCOMES:
Worst-Itch Numeric Rating Scale (WI-NRS-4)-4 at Week 16 | Baseline and Week 16
  Proportion of subjects achieving an improvement of Worst-Itch Numeric Rating Scale (WI-NRS) ≥4 from baseline at Week 16.
Worst-Itch Numeric Rating Scale (WI-NRS-4)-4 at all visits other than Week 16. | Baseline to week 52 other than Week 16.
  Proportion of subjects achieving an improvement of WI-NRS ≥4 from baseline at all scheduled visits other than Week 16.
Change from Baseline in Eczema Area and Severity Index at all visits. | Baseline to week 52
  EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness (erythema, inflammation), thickness (induration, papulation, swelling - acute eczema), scratching (excoriation), and lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease .
Eczema Area and Severity Index (EASI 75) at all visits other than Week 16 | Baseline to week 52 other than Week 16
  Proportion of subjects achieving at least a 75% improvement in Eczema Area and Severity Index (EASI 75) from baseline at all visits other than Week 16.

CONTACTS AND LOCATIONS:
Overall Officials: Jianzhong Zhang, Principal Investigator — Peking University People's Hospital
Locations (1):
- Dermatological Hospital of Southern Medical University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No